CLINICAL TRIAL: NCT00698763
Title: Effects of Oral Levosimendan on Ambulatory Electrocardiographic Variables and Cerebrovascular Reactivity in Patients With Recent Stroke or TIA.
Brief Title: Effects of Oral Levosimendan on Ambulatory Electrocardiographic Variables
Acronym: Electro
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Juha Ellmen, Clinical Program Leader, Orion Pharma
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3001088
Record Dates: First submitted 2008-06-12; First posted 2008-06-17 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2009-11

CONDITIONS: Transient Ischemic Attack; Stroke
Keywords: An ischaemic cerebrovascular event (stroke or TIA)
MeSH Terms: conditions — Ischemic Attack, Transient; Stroke | interventions — Simendan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Levosimendan
  Interventions: Drug: Levosimendan
- B (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levosimendan — from 0.125 mg to 2 mg in escalating doses
  Arms: A
Drug: Placebo — Placebo capsules are identical in appearance to active capsules
  Arms: B

SUMMARY:
The primary objective is to explore the safety of low doses of oral levosimendan in patients with recent history of an ischaemic cerebrovascular event (stroke or TIA). The main focus will be on the evaluation of proarrhythmic potential of the different dose regimens.

DETAILED DESCRIPTION:
This is a prospective, multicentre, phase II, randomized, double-blind, placebo-controlled 2-arm parallel group study with 5 escalating dose-levels of oral levosimendan, each given for 13-18 days. The study population will be randomly allocated either to the levosimendan group or to the placebo group. The double-blind phase with either placebo or levosimendan is preceded by a 13-day long single-blind treatment with placebo (placebo run-in). The study consists of 9 visits (screening visit, 7 visits during the treatment period and an end-of-study visit). Each subject will be on study treatment (including placebo run-in) for 78-108 days and the duration of the study for each subject, including the screening and the end of study visit, is approximately 17 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients 50 to 80 years of age with ischaemic stroke or TIA within 1 to 9 months before the screening visit.

Exclusion Criteria:

* Stroke or TIA due to cardiac embolism, vasculitis or arterial dissection
* Severe hemiparesis or dysphasia, haemodynamically significant uncorrected valve disease or hypertrophic cardiomyopathy or restrictive cardiomyopathy, any acute coronary event or angioplasty or any other major surgery within 1 month, any major surgery during the planned study period
* History of life-threatening ventricular arrhythmia within 3 months.
* History of Torsades de Pointes (TdP) or family history of long QT-syndrome
* Heart rate (HR) < 50 or > 100 bpm.
* Systolic blood pressure (SBP) < 100 mmHg or > 180 mmHg, or diastolic blood pressure (DBP) > 100 mmHg.
* Ventricular tachycardia.
* Episode of atrial fibrillation or atrial flutter lasting > 60 seconds.
* Second or third degree atrioventricular (AV) block.
* Potassium (K) < 3.7 mmol/l or > 5.5 mmol/l.
* Creatinine > 170 µmol/l or on dialysis.
* Blood haemoglobin <10 g/dl; clinically significant hepatic impairment.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-08; Primary Completion 2009-04 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
24-h Holter reporting | every 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Irja Korpela, Study Director — Orion Corporation, Orion Pharma; Risto O. Roine, M.D., Ph.D., Principal Investigator — Turku University Hospital
Locations (7):
- Finland (2):
  - Helsinki University Hospital (HUCH), Helsinki
  - Turku University Hospital (TYKS), Turku
- Heidelberg University Clinic, Heidelberg, Germany
- Debrecen University, Debrecen, Hungary
- Sweden (3):
  - Sahlgrenska University Hospital, Dept of Neurology, Gothenburg
  - University Hospital, Neurologmottagningen, Linköping
  - Umeå University Hospital, Strokecenter NVS, Umeå

REFERENCES:
- [Derived] Kivikko M, Kuoppamaki M, Soinne L, Sundberg S, Pohjanjousi P, Ellmen J, Roine RO. Oral Levosimendan Increases Cerebral Blood Flow Velocities in Patients with a History of Stroke or Transient Ischemic Attack: A Pilot Safety Study. Curr Ther Res Clin Exp. 2015 Jan 29;77:46-51. doi: 10.1016/j.curtheres.2015.01.001. eCollection 2015 Dec. PMID 26082815